CLINICAL TRIAL: NCT05545137
Title: Pivmecillinam Hydrochloride Tablets Versus Fosfomycin Tromethamine Granules for Uncomplicated Urinary Tract Infection in Women -A Randomized, Double-blind, Double Simulation, Positive Drug Parallel-controlled, Multi Center Phase III Clinical Trial in China
Brief Title: Clinical Trial of Pivmecillinam Hydrochloride Tablets in the Treatment of Uncomplicated Urinary Tract Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Benova (Tianjin) Innovative medicine Research Co., Ltd. (Other)
Responsible Party: Sponsor
Organization: Greenpine Pharma Group Co., ltd. (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CS1046
Record Dates: First submitted 2022-09-02; First posted 2022-09-19 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Uncomplicated Urinary Tract Infection
MeSH Terms: interventions — Amdinocillin Pivoxil; Fosfomycin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pivmecillinam hydrochloride tablets treatment group (Experimental): participants received Pivmecillinam Hydrochloride Tablets + Fosfomycin Tromethamine Granules Simulant.
  Pivmecillinam Hydrochloride Tablets:oral,One tablets each time,3 times a day for five days.
  Fosfomycin Tromethamine Granules Simulant :oral, 1 pack, only once for the entire course of treatment
  Interventions: Drug: Pivmecillinam hydrochloride tablets
- Fosfomycin Tromethamine Granules treatment group (Active Comparator): participants received Fosfomycin Tromethamine Granules + Pivmecillinam Hydrochloride Tablets Simulant
  Fosfomycin Tromethamine Granules:oral, 1 pack, only once for the entire course of treatment.
  Pivmecillinam Hydrochloride Tablets Simulant :oral,One tablets each time,3 times a day for five days.
  Interventions: Drug: Fosfomycin Tromethamine Granules

INTERVENTIONS:
Drug: Pivmecillinam hydrochloride tablets — 400mg tablet
  Other Names: Selexid®
  Arms: Pivmecillinam hydrochloride tablets treatment group
Drug: Fosfomycin Tromethamine Granules — 3g/pack
  Other Names: Monurol®
  Arms: Fosfomycin Tromethamine Granules treatment group

SUMMARY:
the purpose of this study is to evaluate the efficacy and safety of pivmecillinam hydrochloride tablets in the treatment of uncomplicated urinary tract infection in China

DETAILED DESCRIPTION:
Screening period (D -3 to D -1): complete screening examinations will be performed after the subject signs the informed consent

Dosing Treatment Period (D 1 to D 5): subjects who met the inclusion criteria and did not meet the exclusion criteria were randomized. Refer to the randomization protocol for specific randomization process.

Safety check (D 5+1): perform on-site visit after 15 doses (D 5+1)

Post-treatment follow-up assessments ((D 12±2) and (D 21+7)): subjects returned to the study site for on-site follow-up on Day 12±2 and Day 21+7.

Urine bacterial culture and minimal inhibitory concentration (MIC) test: urine bacterial culture is required for subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients over 18 years of age with uncomplicated urinary tract infection ;
2. Within 72 hours prior to study entry, the following symptoms or signs occurred: frequency of urine, urgency, dysuria (including suprapubic pain, pain or burning sensation on urination), dysuria, and symptom score ≥ 2 points;
3. Urinalysis showed leukocyturia, i.e.,white blood cells≥ 10/μl on non-centrifuged urinalysis and white blood cell count greater than the upper limit of normal at the study site or white blood cells>5 /HP（high-power） on microscopic examination of urine sediment;
4. Those who have no childbearing plan within the past 6 months (women of childbearing potential have a negative urine pregnancy test result at screening or within 72 hours before starting the trial) and agree to use effective non-drug contraception during the study;
5. Subjects who agree to participate in this clinical trial and sign a written informed consent form (ICF);

Exclusion Criteria:

1. Patients with acute or chronic upper urinary tract infection (eg, temperature > 38 °C, chills, or costovertebral angle pain, etc.);
2. Other factors predisposing to urinary tract infection, including patients with known structural or functional abnormalities of the urinary tract such as urinary calculi;
3. Patients with indwelling catheterization or urinary incontinence;
4. Patients who have taken drugs for treatment of urinary tract infection or antibiotics for other diseases within 48 hours prior to dosing are excluded if the half-life of antibiotics taken by the subject is long and cannot be basically cleared before dosing as judged by the investigator, even if they have not taken any antibiotics within 48 hours prior to randomization;
5. Have taken probenecid, metoclopramide, methotrexate, aspirin, or other antimicrobial agents within 48 hours prior to dosing;
6. Have taken valproic acid or valproic acid-releasing drugs (including sodium valproate, sodium divalproex, etc.) within 48 hours prior to dosing;
7. Previous or current STDs;
8. Previous diabetes mellitus with unregulated treatment showing abnormal blood glucose ;
9. Patients allergic (including lactose intolerance) to penicillins, pivmecillinam, mecillinam, cephalosporins, fosfomycin tromethamine, or other components of the study drug;
10. Patients suspected to be unable to comply with the protocol (e.g., alcoholism, drug dependence, or poor mental status);
11. Patients have been enrolled in this trial;
12. Those who have participated in other drug interventional clinical trials or are participating in other clinical trials within 3 months prior to screening;
13. Patients who have taken study drug within the past 3 months;
14. Pregnant, lactating women, patients who are pregnant during the study or have a fertility plan within 3 months after the end of the trial;
15. Complaints of active gastric ulcer and episodes of hemorrhagic gastritis;
16. Abnormal liver and kidney function tests (ALT, AST ≥ 1.5 times the upper limit of normal, or serum creatinine ≥ 1.5 × upper limit (ULN) or creatinine clearance ≤ 50 mL/min), or other diseases that affect the efficacy of the drug as judged by the investigator ;
17. Those who are judged by the investigator to be ineligible for enrollment by clinical laboratory tests, electrocardiograms, urinary ultrasound, etc.;
18. Other reasons for inappropriate participation in the trial in the opinion of the investigator.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2022-09-29 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Change in urinary tract infection symptom score | From Baseline to Day 12±2
  The Urinary Tract Infection Symptom Score is a validated, self-reported tool to assess the severity of frequency, urgency, pain, dysuria, and may range from 0 (no symptoms) to 12 (worst symptoms).
  Change = (Day 12±2 Score - Baseline Score)
Urine white blood cell count | Day 12±2
  Defined as whether the subject 's white blood cell count returned to normal. The result was yes or no.

SECONDARY OUTCOMES:
Urine culture pathogen count at visit | Day 12±2
  The urine culture pathogenic bacteria count at the visit was defined as: the urine culture pathogen (baseline pathogen) at enrollment was cleared at the visit or the bacterial count was reduced to< 10^3 CFU(Colony-Forming Unit)/ml. The judgment results were: Yes, No, and could not be judged (could not be judged due to lack of culture results).
Change in urinary tract infection symptom score | From Baseline to Day 5+1
  The Urinary Tract Infection Symptom Score is a validated, self-reported tool to assess the severity of frequency, urgency, Urinary pain, dysuria, and may range from 0 (no symptoms) to 12 (worst symptoms).
  Change = (Day 12±2 Score - Baseline Score)
Urine white blood cell count | Day 5+1
  Defined as whether the subject 's white blood cell count returned to normal. The result was yes or no.
Urine culture pathogen count at visit | Day 5+1
  The urine culture pathogenic bacteria count at the visit was defined as: the urine culture pathogen (baseline pathogen) at enrollment was cleared at the visit or the bacterial count was reduced to<10^3 CFU/ml. The judgment results were: Yes, No, and could not be judged (could not be judged due to lack of culture results).
Change in urinary tract infection symptom score | From Baseline to Day 21+7
  The Urinary Tract Infection Symptom Score is a validated, self-reported tool to assess the severity of frequency, urgency, Urinary pain, dysuria, and may range from 0 (no symptoms) to 12 (worst symptoms).
  Change = (Day 12±2 Score - Baseline Score)
Urine white blood cell count | Day 21+7
  Defined as whether the subject 's white blood cell count returned to normal. The result was yes or no.
Urine culture pathogen count at visit | Day 21+7
  The urine culture pathogenic bacteria count at the visit was defined as: the urine culture pathogen (baseline pathogen) at enrollment was cleared at the visit or the bacterial count was reduced to<10^3 CFU/ml. The judgment results were: Yes, No, and could not be judged (could not be judged due to lack of culture results).
Safety variables | Day 5+1,Day 12±2,Day 21+7
  Safety variables: adverse events reported by the patient at the visit or occurred during the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Xiangdong Yang, PhD, Principal Investigator — Qilu Hospital of Shandong University
Locations (10):
- China (10):
  - Beijing hospital, Beijing, Beijing Municipality
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Guangxi Zhuang Autonomous Region People's Hospital, Nanning, Guangxi
  - The second hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Wuhan Central Hospital, Wuhan, Hubei
  - Xiangya Humanity Rehabilitation hospital, Changsha, Hunan
  - Loudi Central Hospital, Loudi, Hunan
  - Yueyang people's Hospital, Yueyang, Hunan
  - Jiangsu Provincial Hospital of Integrated Chinese and Western Medicine, Nanjing, Jiangsu
  - Qilu Hospital of Shandong University, Jinan, Shandong

IPD SHARING:
Plan to Share IPD: No